CLINICAL TRIAL: NCT03458572
Title: Acupuncture for the Prevention of Intrathecal Diamorphine-induced Itch in Elective Caesarean Section: A Randomised Controlled Trial
Brief Title: Acupuncture for Prevention of Itch in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STH20078
Record Dates: First submitted 2018-02-22; First posted 2018-03-08 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pruritus
Keywords: Caesarean section
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1.5mm Seirin Pyonex needle at LI11 point
  Interventions: Device: Seirin Pyonex press needle acupuncture
- Control (Sham Comparator): 0.3mm Seirin Pyonex needle at TB10 point
  Interventions: Device: Seirin Pyonex press needle acupuncture

INTERVENTIONS:
Device: Seirin Pyonex press needle acupuncture — Acupuncture

SUMMARY:
This study aims to determine the effectiveness of using a commercially available acupuncture stud at the LI11 acupuncture point at reducing the severity of itch caused by intrathecal diamorphine in elective caesarean section.

DETAILED DESCRIPTION:
Itch is a very common complication of diamorphine used in spinal anaesthesia for caesarean section with a local incidence of 78%. It ranges from irritating to distressing and difficult to treat and can adversely affect maternal satisfaction, wellbeing and bonding with their baby.

This trial aims to determine whether acupuncture using a commercially-available acupuncture stud at the LI11 point reduces the incidence and severity of post-operative itching in patients undergoing elective caesarean section under spinal anaesthesia with intrathecal diamorphine.

80 women having a planned caesarean section under spinal anaesthesia will be recruited by informed consent and randomised to the intervention group or the control group. The intervention group will receive an acupuncture stud at the LI11 point on either arm and the control group will receive acupuncture with a similar stud containing a smaller needle at a non-acupuncture point on either arm. The stud can be left in-situ until the followup visit the following morning or removed earlier at the participants discretion. All other care will be the usual clinical care including access to anti-itching drugs as required. Participants will be visited by a member of the research team at 3-5 hours following the start of their spinal anaesthetic and asked to mark their itch on an 11 point visual analogue scale (VAS). They will also be visited by a member of the research team the following morning, asked to rate their worst itch on the same scale and asked how troublesome they have found their itch (none, mild, moderate, severe). The administration of any anti-itch drugs will be recorded and if the acupuncture stud has not been removed it will be removed at this time.

If effective, acupuncture with an acupuncture stud would provide an acceptable, convenient, safe and cost-effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* ASA1-3 patients with uncomplicated pregnancies undergoing elective caesarean section with a plan for spinal anaesthesia with intrathecal diamorphine.

Exclusion Criteria:

* Age under 18.
* Pre-existing itch or conditions associated with itch (eg cholestasis of pregnancy).
* Pre-existing use of H1 receptor antagonists, non-selective antihistamines or ursodeoxycholic acid.
* Severe perioperative complication or fetal death.
* Conversion to general anaesthesia.
* Unable to understand written and spoken English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Presence or absence of itch | between 3 and 5 hours post injection of spinal anaesthetic
  Presence or absence of itch

SECONDARY OUTCOMES:
Severity of itch on 11 point VAS scale | between 3 and 5 hours post injection of spinal anaesthetic
  Severity of itch on 11 point VAS scale
Severity of worst overall itch on 11 point VAS scale | At a follow up visit the next day following the spinal anaesthetic
  Severity of worst overall itch on 11 point VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Tim Orr, Dr, Principal Investigator — Trainee Anaesthesia (CT1-ST6)
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No